CLINICAL TRIAL: NCT03086486
Title: A Phase 3 Partially-blinded, Randomized Trial Assessing the Safety and Efficacy of Various Doses and Treatment Durations of Linezolid Plus Bedaquiline and Pretomanid in Participants With Pulmonary Infection of Either Extensively Drug-resistant Tuberculosis (XDR-TB), Pre-XDR-TB or Treatment Intolerant or Non-responsive Multi-drug Resistant Tuberculosis (MDR-TB)
Brief Title: Various Doses and Durations of Linezolid Plus Bedaquiline & Pretomanid in Participants With Drug Resistant Tuberculosis
Acronym: ZeNix
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Global Alliance for TB Drug Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZeNix (B-Pa-L) NC-007
Record Dates: First submitted 2017-03-07; First posted 2017-03-22 (Actual); Results first posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Tuberculosis, Pulmonary; Tuberculosis, Multidrug-Resistant; Tuberculosis, MDR; Tuberculosis; Extensively Drug-Resistant Tuberculosis; Pre-XDR-TB; XDR-TB
Keywords: Tuberculosis; Multi Drug-Resistant Tuberculosis; Extensively Drug-Resistant Tuberculosis; Drug-Resistant Tuberculosis; Pretomanid; PA-824; Bedaquiline; Linezolid; NC-007; TB Alliance; pre-XDR-TB; Sirturo; Zyvox; ZeNix
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis, Multidrug-Resistant; Tuberculosis; Extensively Drug-Resistant Tuberculosis | interventions — pretomanid; Linezolid; bedaquiline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants, trial investigators and staff, including laboratory staff, will be blinded to dose and scheduled duration of linezolid. Bedaquiline and pretomanid dosing will not be blinded. There will be three unblinded analyses which will contain results by linezolid treatment group in aggregate. The first analysis will be after all participants have completed 26 weeks of treatment and here sites, participants, and Sponsor staff will not be unblinded to individual linezolid treatment information. A limited number of statisticians will have access to individual linezolid treatment assignments. The blind for all individual participants will be broken for the primary endpoint analysis (the second unblinded analysis) once all clinical data and outcome parameters have been captured, no more data queries are pending, and the statistical analysis plan has been finalized. The third analysis will occur when all participants have completed 78 weeks of follow-up after end of treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 1200mg L x 26 weeks + Pa + B (Experimental): 2 linezolid 600 mg active tablets once daily for 26 weeks plus 1 placebo linezolid 300 mg half tablet once daily for 26 weeks plus; bedaquiline 200 mg once daily for 8 weeks then 100 mg once daily for 18 weeks plus; pretomanid 200 mg once daily for 26 weeks
  Interventions: Drug: Pretomanid; Drug: Linezolid; Drug: Bedaquiline; Drug: Placebo Linezolid
- 1200 mg L x 9 weeks + Pa + B (Experimental): 2 linezolid 600 mg active tablets once daily for 9 weeks, 1 placebo linezolid 300 mg half tablet once daily for 9 weeks (for Weeks 1-9); 2 placebo linezolid 600 mg tablets once daily for 17 weeks, 1 placebo linezolid 300 mg half tablet once daily for 17 weeks (for Weeks 10-26) plus; bedaquiline 200 mg once daily for 8 weeks then 100 mg once daily for 18 weeks plus; pretomanid 200 mg once daily for 26 weeks
  Interventions: Drug: Pretomanid; Drug: Linezolid; Drug: Bedaquiline; Drug: Placebo Linezolid
- 600 mg L x 26 weeks + Pa + B (Experimental): 1 linezolid 600 mg active tablet once daily for 26 weeks, 1 placebo linezolid 600 mg tablet once daily for 26 weeks, 1 placebo linezolid 300 mg half tablet once daily for 26 weeks plus; bedaquiline 200 mg once daily for 8 weeks then 100 mg once daily for 18 weeks plus; pretomanid 200 mg once daily for 26 weeks
  Interventions: Drug: Pretomanid; Drug: Linezolid; Drug: Bedaquiline; Drug: Placebo Linezolid
- 600 mg L x 9 weeks + Pa + B (Experimental): 1 linezolid 600 mg active tablets once daily for 8 weeks, 1 placebo linezolid 600 mg half tablet once daily for 9 weeks, 1 placebo linezolid 300 mg half tablet once daily for 9 weeks (for Weeks 1-9); 2 placebo linezolid 600 mg tablets once daily for 17 weeks, 1 placebo linezolid 300 mg half tablet once daily for 17 weeks (for Weeks 10-26) plus; bedaquiline 200 mg once daily for 8 weeks then 100 mg once daily for 18 weeks plus; pretomanid 200 mg once daily for 26 weeks
  Interventions: Drug: Pretomanid; Drug: Linezolid; Drug: Bedaquiline; Drug: Placebo Linezolid

INTERVENTIONS:
Drug: Pretomanid — 200mg tablets
  Other Names: PA-824; Pa
Drug: Linezolid — Scored 600mg tablets
  Other Names: L; Lin; Zyvox
Drug: Bedaquiline — 100mg tablets
  Other Names: TMC-207; B; Sirturo
Drug: Placebo Linezolid — Scored 600 mg tablets

SUMMARY:
To evaluate the efficacy, safety and tolerability of various doses and durations of linezolid plus bedaquiline and pretomanid after 26 weeks of treatment in participants with either pulmonary XDR-TB, pre-XDR-TB, or treatment intolerant or non-responsive MDR-TB.

DETAILED DESCRIPTION:
A phase 3, multi-center, partially-blinded, randomized clinical trial in 4 parallel treatment groups. Bedaquiline and pretomanid treatment will not be blinded. Linezolid treatment dose and duration will be double-blinded.

Participants will have a screening period of up to 14 days and will be randomized to receive one of the 4 active treatment arms. Participants will be randomized to one of the 4 regimens in a 1:1:1:1 ratio, using an interactive voice and web response system (IXRS) which will utilize a randomization system using stratification with a random element to allocate participants evenly across the arms by HIV status and type of TB.

Each participant will receive 26 weeks of treatment. If participant's week 16 sputum sample is culture positive between the week 16 and week 26 treatment visits and their clinical condition suggests they may have an ongoing TB infection, Investigator may consider extending current treatment to 39 weeks. If the culture results between week 16 and week 26 are contaminated, missing or considered an isolated positive without clinical significance, available culture results should be used to make this decision. All decisions regarding treatment extension should be discussed with and approved by, in consultation with the Sponsor Medical Monitor before implementation. The treatment may also require modification due to toxicities. All dose modifications should be discussed with the Sponsor Medical Monitor prior to implementation, unless a pause or dose reduction is required urgently for safety concerns.

Participants will be followed for 78 weeks after end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 14 years or older.
* One of the following with documentation of culture positive or molecular test within 3 months of screening:

  * XDR-TB defined as resistance to rifamycins, a fluoroquinolone AND an injectable OR
  * Pre-XDR-TB with defined as resistance to rifamycins, and to a fluoroquinolone OR an injectable OR
  * MDR-TB with resistance to rifamycins, and either non-responsive or non-tolerant to current treatment.
* Of non-childbearing potential or willing to practice effective birth control methods.
* Complete informed consent form.

Exclusion criteria:

* Karnofsky score < 60 at screening.
* Body mass index (BMI) < 17 kg/m2
* Participants who are expected to require a surgical procedure (for Pulmonary TB).
* Any risk factor for QT prolongation
* Pregnant or breast-feeding
* Any planned contraindicated medicines or received more than 2 weeks of bedaquiline, linezolid or delamanid prior to first dose of IMP.
* A peripheral neuropathy of Grade 3 or 4, according to DMID. Or, participants with a Grade 1 or 2 neuropathy which is likely to progress/worsen over the course of the study, in the opinion of the Investigator
* Any of the following lab toxicities/abnormalities:

  * Viral load >1000 copies/mL (Unless newly diagnosed HIV and not yet on ART who otherwise qualify for participation);
  * CD4+ count < 100 cells/µL (HIV positive participants);
  * Serum potassium less than the lower limit of normal for the laboratory;
  * Hemoglobin < 9.0 g/dL or 90g/L;
  * Platelets <100,000/mm3 or < 100 x 10^9/L
  * Absolute neutrophil count (ANC) < 1500/ mm3 or < 1.5 x 10^9/L
  * Aspartate aminotransferase (AST) and Alanini aminotransferase (ALT) Grade 3 or greater (> 3.0 x ULN)
  * Total bilirubin greater than 1.5 x ULN
  * Direct bilirubin greater than ULN
  * Serum creatinine level greater than 1.5 times upper limit of normal
  * Albumin <3.0 g/dl or < 30 g/L

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2022-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Conradie, Principal Investigator — Isango Lethemba TB Research Unit
Locations (11):
- National Center for Tuberculosis and Lung Diseases, Tbilisi, Georgia
- Institute of Phthisiopneumology Chiril Draganiuc, Chisinau, Moldova
- Russia (5):
  - Moscow City Research and Practice Tuberculosis Treatment Centre, Moscow
  - Central TB Research Institute of the Federal Agency of Scientific Organizations Moscow, Moscow
  - National Medical Research Center of Phthisiopulmonology and Infectious Diseases, Moscow
  - FSBI "Saint-Petersburg Research Institute of Phthisiopulmonology", Saint Petersburg
  - Ural Research Institute of Phthisiopulmonology, Yekaterinburg
- South Africa (4):
  - Empilweni TB Hospital, Port Elizabeth, Eastern Cape
  - Tshepong Hospital, Klerksdorp, North West
  - King DinuZulu Hospital Complex, Durban
  - Clinical HIV Research Unit (CHRU) Sizwe Tropical Diseases Hospital, Johannesburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Conradie F, Bagdasaryan TR, Borisov S, Howell P, Mikiashvili L, Ngubane N, Samoilova A, Skornykova S, Tudor E, Variava E, Yablonskiy P, Everitt D, Wills GH, Sun E, Olugbosi M, Egizi E, Li M, Holsta A, Timm J, Bateson A, Crook AM, Fabiane SM, Hunt R, McHugh TD, Tweed CD, Foraida S, Mendel CM, Spigelman M; ZeNix Trial Team. Bedaquiline-Pretomanid-Linezolid Regimens for Drug-Resistant Tuberculosis. N Engl J Med. 2022 Sep 1;387(9):810-823. doi: 10.1056/NEJMoa2119430. PMID 36053506

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 248 participants were screened for the trial, of whom 67 failed screening, 181 were randomized, and 169 completed treatment.
Period: Overall Study
Arm/Group | 1200mg L x 26 Weeks + Pa + B | 1200 mg L x 9 Weeks + Pa + B | 600 mg L x 26 Weeks + Pa + B | 600 mg L x 9 Weeks + Pa + B
Started | 45 | 46 | 45 | 45
Completed (Treatment) | 44 | 42 | 43 | 40
Not Completed | 1 | 4 | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1200mg L x 26 Weeks + Pa + B | 1200 mg L x 9 Weeks + Pa + B | 600 mg L x 26 Weeks + Pa + B | 600 mg L x 9 Weeks + Pa + B | Total
Number analyzed (Participants) | 45 | 46 | 45 | 45 | 181
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 37.4 [30.0 to 44.0] | 35.1 [26.0 to 42.0] | 39.2 [30.0 to 46.0] | 36.8 [32.0 to 41.0] | 37.1 [30.0 to 44.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 14 | 14 | 59
  Male | 30 | 30 | 31 | 31 | 122
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 11 | 18 | 21 | 16 | 66
  White | 34 | 28 | 24 | 29 | 115
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 11 | 18 | 21 | 16 | 66
  Moldova | 2 | 4 | 1 | 3 | 10
  Georgia | 13 | 8 | 5 | 8 | 34
  Russia | 19 | 16 | 18 | 18 | 71
Height [Mean (Inter-Quartile Range); unit: cm] | 173.2 [165.0 to 178.0] | 170.2 [164.0 to 177.0] | 171.2 [165.0 to 174.0] | 171.2 [164.0 to 179.0] | 171.4 [165.0 to 178.0]
Weight [Mean (Inter-Quartile Range); unit: kg] | 62.8 [55.0 to 67.3] | 62.1 [52.9 to 69.0] | 63.1 [52.4 to 66.5] | 64.5 [58.0 to 70.7] | 63.1 [54.0 to 67.8]
BMI [Mean (Inter-Quartile Range); unit: kg/m^2] | 20.8 [18.8 to 22.3] | 21.3 [18.6 to 23.4] | 21.3 [18.6 to 23.6] | 21.9 [19.6 to 24.0] | 21.3 [18.8 to 23.2]
HIV Status [Count of Participants; unit: Participants]
  Positive | 9 | 9 | 9 | 9 | 36
  Negative | 36 | 37 | 36 | 36 | 145
Smoking [Count of Participants; unit: Participants]
  Never | 20 | 15 | 16 | 17 | 68
  Current | 15 | 22 | 17 | 12 | 66
  Former | 10 | 9 | 12 | 16 | 47
Alcohol Use [Count of Participants; unit: Participants]
  Never | 21 | 13 | 18 | 11 | 63
  Current | 8 | 8 | 8 | 10 | 34
  Former | 16 | 25 | 19 | 24 | 84
Karnofsky performance status [Count of Participants; unit: Participants] — Trained clinicians interview participants and grade their ability to perform daily activities using a percent scale where higher scores indicate that the participant is better able to function than lower scores. 100% indicates normal activity with no evidence of disease whereas a score of 70% or lower would indicate that the participant is unable to work and 40% or lower is unable to care for themselves. http://www.npcrc.org/files/news/karnofsky_performance_scale.pdf
  Participants
    100 | 1 | 1 | 2 | 4 | 8
    90 | 28 | 30 | 29 | 26 | 113
    80 | 13 | 13 | 10 | 11 | 47
    70 | 3 | 2 | 4 | 4 | 13
    60 or below | 0 | 0 | 0 | 0 | 0
Current Tuberculosis (TB) type [Count of Participants; unit: Participants]
  Multi Drug Resistant (MDR) TB (nonresponsive) | 2 | 5 | 2 | 3 | 12
  Multi Drug Resistant (MDR) TB (treatment-intolerant) | 3 | 1 | 2 | 3 | 9
  Pre-Extensively Drug Resistant (Pre-XDR) TB | 19 | 22 | 22 | 22 | 85
  Extensively Drug Resistant (XDR) TB | 21 | 18 | 19 | 17 | 75
History of Tuberculosis (TB) [Number; unit: participants] — Participants reported all previous tuberculosis infections prior to and including current infection.
  participants
    Drug Sensitive (DS) TB | 16 | 13 | 18 | 7 | 54
    Mono Resistant TB | 0 | 0 | 1 | 1 | 2
    MDR TB | 20 | 23 | 21 | 25 | 89
    Pre-XDR TB | 6 | 5 | 6 | 7 | 24
    XDR TB | 25 | 28 | 28 | 25 | 106
Screening smear microscopy for Acid Fast Bacilli (AFB) [Count of Participants; unit: Participants] — Detected acid-fast bacilli (AFB) by microscopic examination of clinical sputum specimens and cultures collected from participants. A quantitative grading system (WHO/IUATLD scaling system) was used to report the number of AFB observed in stained smears from concentrated sputum specimens, ranging from none seen to a 3+, depending on the amount of bacilli counted on microscopic examination.
  Participants
    No AFB seen | 23 | 24 | 23 | 20 | 90
    Scanty positive | 11 | 4 | 8 | 5 | 28
    1+ | 4 | 7 | 4 | 6 | 21
    2+ | 6 | 6 | 3 | 4 | 19
    3+ | 1 | 5 | 7 | 10 | 23
Time to positive at baseline [Mean (Inter-Quartile Range); unit: days] — Liquid culture in the MGIT platform to detect the presence or absence of Mycobacterium tuberculosis (MTB) and obtain the time to positivity (TTP) Population: Only participants who were positive at baseline in liquid culture MGIT. Positive culture at screening not required per protocol.
  days
    number analyzed (Participants) | 30 | 32 | 33 | 36 | 131
    (all) | 14.3 [6.9 to 16.8] | 11.3 [6.7 to 13.7] | 14.0 [5.7 to 20.3] | 12.5 [5.8 to 17.7] | 13.0 [6.5 to 16.8]
Chest x-ray at Screening [Count of Participants; unit: Participants] — Obtained and read locally by the investigator or designee with results classified as normal or abnormal consistent with pulmonary TB in the opinion of the investigator.
  Participants
    Normal | 2 | 2 | 1 | 2 | 7
    Abnormal | 43 | 44 | 44 | 43 | 174
Chest X-ray Cavities at Screening [Count of Participants; unit: Participants]
  None | 18 | 21 | 12 | 18 | 69
  Unilateral | 22 | 21 | 20 | 21 | 84
  Bilateral | 5 | 4 | 13 | 6 | 28

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Bacteriologic Failure or Relapse or Clinical Failure (Unfavorables) Through Follow up Until 26 Weeks After the End of Treatment
Description: Unfavourable status:
  1. Participants not classified as having achieved or maintained culture negative status when last seen
  2. Participants previously classified as having culture negative status who, following the end of treatment, have two positive cultures without an intervening negative culture
  3. Participants who had a positive culture not followed by at least two negative cultures when last seen
  4. Participants dying from any cause during treatment, except from violent or accidental cause, not including suicide
  5. Participants definitely or possibly dying from TB related cause during the follow-up phase
  6. Participants requiring an extension of their treatment beyond that permitted by the protocol a restart or a change of treatment for any reason except reinfection or pregnancy
  7. Participants who have had surgery and the resected tissue is cultured and is positive for MTB
  8. Participants lost to follow up or withdrawn from the study before the end of treatment
Time Frame: 26 weeks
Population: Participants were considered unassessable and therefore excluded from the Modified Intent to Treat (MITT) population if they were late exclusions, lost to follow-up, reinfected with a different strain of TB, withdrawn during the Follow-up Period, or died during the treatment period.
Measure: Count of Participants; unit: Participants
Groups:
- Total: Total Study Population
Arm/Group | 1200mg L x 26 Weeks + Pa + B | 1200 mg L x 9 Weeks + Pa + B | 600 mg L x 26 Weeks + Pa + B | 600 mg L x 9 Weeks + Pa + B | Total
Number analyzed (Participants) | 44 | 45 | 45 | 44 | 178
Participants
  Favorable | 41 | 40 | 41 | 37 | 159
  Unfavorable | 3 | 5 | 4 | 7 | 19

2. Secondary Outcome: Incidence of Bacteriologic Failure or Relapse or Clinical Failure (Unfavorables) Through Follow up Until 78 Weeks After the End of Treatment.
Description: as for outcome 1
Time Frame: 78 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 1200mg L x 26 Weeks + Pa + B | 1200 mg L x 9 Weeks + Pa + B | 600 mg L x 26 Weeks + Pa + B | 600 mg L x 9 Weeks + Pa + B | Total
Number analyzed (Participants) | 43 | 44 | 45 | 44 | 176
Participants
  Favorable | 40 | 39 | 40 | 35 | 154
  Unfavorable | 3 | 5 | 5 | 9 | 22

3. Secondary Outcome: Time to Sputum Culture Conversion to Negative Status Through the Treatment Period
Description: Culture conversion is a diagnostic criteria indicating the point at which samples taken from a patient infected with tuberculosis can no longer produce tuberculosis cell cultures.
  Note:
  * Culture conversion requires at least 2 consecutive culture negative/positive samples at least 7 days apart.
  * Participants who are documented at a visit as unable to produce sputum and who are clinically considered to be responding well to treatment will be considered to be culture negative at that visit.
Time Frame: 26 weeks
Population: Participants in the MITT population who were culture positive during the baseline period were assessable. Unassessable Includes participants not positive at baseline and/or unassessable in the MITT population.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | 1200mg L x 26 Weeks + Pa + B | 1200 mg L x 9 Weeks + Pa + B | 600 mg L x 26 Weeks + Pa + B | 600 mg L x 9 Weeks + Pa + B | Total
Number analyzed (Participants) | 30 | 32 | 33 | 35 | 130
weeks | 4 [2 to 8] | 4 [2 to 8] | 6 [3 to 6] | 6 [3 to 10] | 6 [3 to 8]

4. Secondary Outcome: Sputum Culture Conversion to Negative Status at End of Treatment for Those Positive at Baseline
Description: Culture conversion is a diagnostic criteria indicating the point at which samples taken from a patient infected with tuberculosis can no longer produce tuberculosis cell cultures.
Time Frame: End of Treatment, 26 weeks
Population: The participant numbers for inclusion in analysis are those assessable participants with a positive culture status at baseline, not including those who withdrew or were lost to contact during treatment at or before Week 26.
Measure: Count of Participants; unit: Participants
Arm/Group | 1200mg L x 26 Weeks + Pa + B | 1200 mg L x 9 Weeks + Pa + B | 600 mg L x 26 Weeks + Pa + B | 600 mg L x 9 Weeks + Pa + B | Total
Number analyzed (Participants) | 29 | 29 | 32 | 32 | 122
Participants
  Negative | 29 | 28 | 31 | 31 | 119
  Positive | 0 | 1 | 1 | 1 | 3
  Died | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 28 weeks
Description: All listed adverse events (AEs) are treatment emergent adverse events (TEAE) which are defined as AEs that started or worsened at or after the first administration of IMP up to and including 14 days after the last administration of IMP.
Arm/Group | 1200mg L x 26 Weeks + Pa + B | 1200 mg L x 9 Weeks + Pa + B | 600 mg L x 26 Weeks + Pa + B | 600 mg L x 9 Weeks + Pa + B | Total
All-Cause Mortality (participants affected / at risk) | 0/45 | 1/46 | 0/45 | 0/45 | 1/181
Serious Adverse Events (participants affected / at risk) | 3/45 | 4/46 | 1/45 | 3/45 | 11/181
Other Adverse Events (participants affected / at risk) | 40/45 | 41/46 | 39/45 | 36/45 | 156/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1200mg L x 26 Weeks + Pa + B (N=45) | 1200 mg L x 9 Weeks + Pa + B (N=46) | 600 mg L x 26 Weeks + Pa + B (N=45) | 600 mg L x 9 Weeks + Pa + B (N=45) | Total (N=181)
Optic neuropathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Hepatitis B (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tertiary syphilis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Optic neuritis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alcoholic psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1200mg L x 26 Weeks + Pa + B (N=45) | 1200 mg L x 9 Weeks + Pa + B (N=46) | 600 mg L x 26 Weeks + Pa + B (N=45) | 600 mg L x 9 Weeks + Pa + B (N=45) | Total (N=181)
Anaemia (Blood and lymphatic system disorders) | 7 | 3 | 1 | 3 | 14
Neutropenia (Blood and lymphatic system disorders) | 3 | 6 | 3 | 4 | 16
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 1 | 5 | 12
Dyspepsia (Gastrointestinal disorders) | 4 | 3 | 1 | 1 | 9
Nausea (Gastrointestinal disorders) | 6 | 5 | 1 | 3 | 15
Vomiting (Gastrointestinal disorders) | 3 | 3 | 1 | 2 | 9
Upper respiratory tract infection (Infections and infestations) | 1 | 4 | 2 | 2 | 9
Hepatic enzyme increased (Investigations) | 5 | 8 | 4 | 3 | 20
Transaminases increased (Investigations) | 2 | 3 | 6 | 5 | 16
Headache (Nervous system disorders) | 4 | 5 | 1 | 3 | 13
Hypoaesthesia (Nervous system disorders) | 4 | 4 | 5 | 1 | 14
Paraesthesia (Nervous system disorders) | 2 | 3 | 3 | 3 | 11
Peripheral sensory neuropathy (Nervous system disorders) | 9 | 6 | 4 | 2 | 21
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 3 | 5 | 3 | 13
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 3 | 3 | 10
Rash papular (Skin and subcutaneous tissue disorders) | 3 | 4 | 1 | 2 | 10
Hypertension (Vascular disorders) | 5 | 1 | 2 | 4 | 12

LIMITATIONS AND CAVEATS:
None reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and Principal Investigator shall not publish, present or use the Study Data for its own instruction, research or publication without the prior express written consent of Sponsor. Because the Study is funded, in whole or in part, by the Bill and Melinda Gates Foundation (the "Foundation"), all peer-reviewed published research relating to the Study must comply with the Foundation's Open Access Policy.

DOCUMENTS (3):
  • Study Protocol (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/86/NCT03086486/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-29): https://cdn.clinicaltrials.gov/large-docs/86/NCT03086486/SAP_001.pdf
  • Informed Consent Form (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/86/NCT03086486/ICF_002.pdf